CLINICAL TRIAL: NCT04922697
Title: Reducing PM2.5 Exposure and Lung Cancer Risk Using Spatial Data Science (The Air Study)
Brief Title: Educational Intervention for the Promotion of Knowledge and Preventive Health Behaviors Related to Personal Air Pollution Exposure, The Air Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: Prevent Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RG1121435; NCI-2021-04399 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10685 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2021-06-01; First posted 2021-06-11 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prevention (educational videos, questionnaires) (Experimental): Participants watch 2 educational videos during week 3 regarding air pollution, health effects, and personal preventive health behaviors to reduce air pollution exposure. Participants will use wearable air pollution sensors. Participants will complete questionnaires at weeks 1 and 5.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Watch educational videos and use wearable air pollution sensor
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This clinical trial will conduct an educational intervention to promote knowledge of and preventive health behaviors related to personal air pollution exposure. Air pollution is n ubiquitous environmental exposure that is associated with harmful health effects including lung cancer. The educational intervention is comprised of 2 educational videos that include information regarding air pollution, health effects, and personal preventive health behaviors to reduce air pollution exposure and the use of a wearable air pollution sensor. The knowledge gained from this study may inform future research that will be designed to promote awareness of air pollution and its health effects.

DETAILED DESCRIPTION:
OUTLINE:

Participants watch 2 educational videos during week 3 regarding air pollution, health effects, and personal preventive health behaviors to reduce air pollution exposure. Participants complete questionnaires at weeks 1 and 5.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older: The evidence for personal strategies to reduce air pollution exposure has been focused on adults
* Live in Seattle, WA: The study is designed to focus on Seattle, WA such as using EnviroFlash alerts
* Own a smartphone: The participant requires a smartphone to setup the Flow app for the air pollution sensor
* Not traveling in the near-term: The study is designed to assess air pollution patterns in the local Seattle area
* Leave your home for at least 7 hours per week: Participants will use a wearable air pollution sensor to measure air pollutant levels from indoor and outdoor sources

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-03-05 (Actual)

PRIMARY OUTCOMES:
Changes in knowledge regarding air pollution | At baseline and week 5
  Will calculate the proportion of the items that were answered correctly. McNemar's tests will be used to calculate differences in the proportion of participants answering air pollution knowledge items correctly at baseline and at week 5.
Changes in air pollution preventive health behaviors | At baseline and week 5
  Will calculate summary scores for air pollution preventive health behaviors and paired t-test to determine intervention effectiveness at baseline and at week 5.

SECONDARY OUTCOMES:
Changes in perceived barriers | At baseline and week 5
  Summary scores for perceived barriers (guided by the Health Belief Model) will be calculated from participant questionnaire responses by summing the scores across the relevant scale. Paired t-tests will determine changes in perceived barriers at baseline and week 5.
Changes in perceived benefits | At baseline and week 5
  Summary scores for perceived benefits (guided by the Health Belief Model) will be calculated from participant questionnaire responses by summing the scores across the relevant scale. Paired t-tests will determine changes in perceived benefits at baseline and week 5.
Changes in perceived susceptibility | At baseline and week 5
  Summary scores for perceived susceptibility (guided by the Health Belief Model) will be calculated from participant questionnaire responses by summing the scores across the relevant scale. Paired t-tests will determine changes in perceived susceptibility at baseline and week 5.
Changes in perceived severity | At baseline and week 5
  Summary scores for perceived severity (guided by the Health Belief Model) will be calculated from participant questionnaire responses by summing the scores across the relevant scale. Paired t-tests will determine changes in perceived severity at baseline and week 5.
Changes in self-efficacy | At baseline and week 5
  Summary scores for self-efficacy (guided by the Health Belief Model) will be calculated from participant questionnaire responses by summing the scores across the relevant scale. Paired t-tests will determine changes in self-efficacy at baseline and week 5.
Changes in cues to action | At baseline and week 5
  Will calculate frequencies for each cue to action (guided by the Health Belief Model). McNemar's tests will be used to calculate differences in the proportion of participants regarding each cue to action at baseline and week 5.
Changes in air pollutant levels measured using the Flow 2 personal air quality sensor | At baseline and week 2 vs. week 4 and week 5
  Paired t-tests will determine changes in air pollutant levels at baseline and week 2 vs. week 4 and week 5.
Intervention feasibility (accessibility) | At week 5
  Will report descriptive statistics for intervention accessibility based on responses to the relevant questionnaire items at week 5.
Intervention feasibility (acceptability) | At week 5
  Will report descriptive statistics for intervention acceptability based on responses to the relevant questionnaire items at week 5.
Intervention feasibility (demand) | At week 5
  Will report descriptive statistics for intervention demand based on responses to the relevant questionnaire items at week 5.
Intervention feasibility (uptake, sensor upload completion) | At baseline through week 5
  Will report descriptive statistics the proportion of participants completing sensor uploads.
Intervention feasibility (uptake, educational video viewing) | At week 3
  Will report descriptive statistics for the proportion of viewing educational videos at week 3.
Intervention feasibility (uptake, questionnaire completion) | At baseline and week 5
  Will report descriptive statistics for the proportion of completing the questionnaires at baseline and week 5.

CONTACTS AND LOCATIONS:
Overall Officials: Trang VoPham, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/97/NCT04922697/ICF_000.pdf